CLINICAL TRIAL: NCT01482663
Title: Chronic Hand Eczema - Self-management and Prognosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Gentofte, Copenhagen (Other)
Collaborators: TrygFonden, Denmark (Industry)
Responsible Party: Principal Investigator, Annette Mollerup, MScHealth, PhD-student, University Hospital, Gentofte, Copenhagen
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CHE-2011-Geh
Record Dates: First submitted 2011-11-23; First posted 2011-11-30 (Estimated); Last update posted 2014-12-03 (Estimated); Status verified 2014-12

CONDITIONS: Chronic Hand Eczema; Chronic Hand Dermatitis
Keywords: Hand eczema; Hand dermatitis; Chronic hand eczema; Chronic hand dermatitis; Contact dermatitis; Skin disease; Self-management
MeSH Terms: conditions — Dermatitis, Contact; Skin Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Chronic hand eczema patients (No Intervention): Written information sheets and a 14-minutes DVD about hand eczema handed out by the dermatologist
- Behavioral: Healthy Skin Clinic (Experimental): 1-2 counselling sessions with a nurse, tailored according to individual risks and resources and user access to a website comprising a self-monitoring log, a patients' forum and the possibility of communication with the intervention team of nurses
  Interventions: Behavioral: Healthy Skin Clinic

INTERVENTIONS:
Behavioral: Healthy Skin Clinic — The intervention is founded upon three concurrent elements. Firstly, a SKIN-profile generated by data from a baseline questionnaire (S=Susceptibility, K=Competencies, I=Individual characteristics, N=Necessary precautions).
  Secondly, a patient self-management book which includes a patient's log and is offered in both an online and a physical form. Also support to self-management is offered through possible asynchronous communication and networking.
  Finally, a counselling consultation with a nurse, trained within dermatology.
  Arms: Behavioral: Healthy Skin Clinic

SUMMARY:
Hand eczema is a common disease which often gives a chronic course thus affecting many functions in daily life. The body of evidence related to self-management of chronic hand eczema is poor. Better methods to support self-management of patients with chronic hand eczema may potentially improve the prognosis of a disease which is both a tremendous burden to the individual and to the society. The purpose of this trial is to evaluate the effect of a newly designed guidance programme offering individual counselling compared to conventional information with written information sheets.

DETAILED DESCRIPTION:
Detailed description of the trial and the intervention can be found in the publication:

Mollerup A, Veien NK, Johansen JD. Chronic hand eczema--self-management and prognosis: a study protocol for a randomised clinical trial'. BMC Dermatol. 2012 Jun 12;12:6. doi: 10.1186/1471-5945-12-6.

PMID: 22691871 [PubMed - indexed for MEDLINE] Free PMC Article

ELIGIBILITY:
Inclusion Criteria:

* Patients clinically diagnosed with hand eczema at the first medical consultation at the outpatient ward, Copenhagen University Hospital Gentofte or at a private dermatologic practise in Aalborg, Denmark
* Patients who have given a signed informed consent to participate

Exclusion Criteria:

* Patients who cannot reply to a questionnaire in Danish

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 306 (Actual)
Dates: Start 2011-05; Primary Completion 2012-11 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Hand Eczema Severity Index (HECSI) | 6 months
  Objective assessment of disease severity, measured by HECSI-score at time = 6 months versus HECSI-score at time = 0.

SECONDARY OUTCOMES:
Dermatology Life Quality Index (DLQI) | 6 months
  DLQI measured by questionnaire at time = 6 months versus DLQI measured by questionnaire at time = 0.
Overall burden of disease (VAS) | 6 months
  VAS measured by questionnaire at time = 6 months versus VAS measured by questionnaire at time = 0.
Danish version of The Medication Adherence Report Scale (DMARS-4) | 6 months
  DMARS-4 measured by questionnaire at time = 6 months versus DMARS-4 measured by questionnaire at time = 0 months.

CONTACTS AND LOCATIONS:
Overall Officials: Annette Mollerup, MScHealth, Principal Investigator — University Hospital, Gentofte, Copenhagen; Jeanne D Johansen, Prof, DMSc, Study Director — University Hospital, Gentofte, Copenhagen
Locations (2):
- Denmark (2):
  - Dermatologic practise, Vesterbro 99, Aalborg
  - Department of Dermato-Allergology, Copenhagen University Hospital Gentofte, Hellerup

REFERENCES:
- [Result] Mollerup A, Veien NK, Johansen JD. Effectiveness of the Healthy Skin Clinic--a randomized clinical trial of nurse-led patient counselling in hand eczema. Contact Dermatitis. 2014 Oct;71(4):202-14. doi: 10.1111/cod.12243. Epub 2014 Apr 25. PMID 24766387
- [Result] Mollerup A, Veien NK, Johansen JD. An analysis of gender differences in patients with hand eczema - everyday exposures, severity, and consequences. Contact Dermatitis. 2014 Jul;71(1):21-30. doi: 10.1111/cod.12206. Epub 2014 Mar 12. PMID 24618009
- [Derived] Mollerup A, Veien NK, Johansen JD. Chronic hand eczema--self-management and prognosis: a study protocol for a randomised clinical trial. BMC Dermatol. 2012 Jun 12;12:6. doi: 10.1186/1471-5945-12-6. PMID 22691871